CLINICAL TRIAL: NCT00129506
Title: Comparing Methotrexate Followed by Misoprostol to Misoprostol Alone for Early Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wiebe, Ellen, M.D. (Other)
Collaborators: Ibis Reproductive Health (Other)
Responsible Party: Principal Investigator, Ellen R Wiebe, MD, Principal Investigator, Wiebe, Ellen, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: c04-0636
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Unwanted Pregnancies
Keywords: medical abortion; methotrexate; misoprostol
MeSH Terms: interventions — Methotrexate; Misoprostol

INTERVENTIONS:
Drug: methotrexate + misoprostol
Drug: misoprostol

SUMMARY:
Background: In most countries in which abortion is legal, medical abortions are induced with mifepristone and misoprostol. Since mifepristone is expensive and unavailable in many countries, it is important to find other regimens. Methotrexate, which is used with misoprostol in Canada, is also difficult to obtain in many countries. Misoprostol is inexpensive and available in almost all countries. A report from Nigeria found that 98% of 100 women aborted within 24 hours of using misoprostol given both sublingually and vaginally.

Method: This will be a randomized controlled trial of the usual regimen used in Canada, methotrexate 50 mg/m2 intramuscularly (IM) followed three days later by 800 mcg vaginal misoprostol to the Nigerian regimen of 400 mcg sublingual misoprostol with 400 mcg vaginal misoprostol. The main outcome measure will be a completed abortion within the first week with secondary outcome measures including total surgery rate, time to abortion, complications, pain, side effects and patient satisfaction.

Rationale: If the investigators can find an inexpensive, easily available, method of medical abortion, it will save many lives in third world countries.

DETAILED DESCRIPTION:
Background/Rationale:

Medical abortions induced with either mifepristone or methotrexate and then followed by misoprostol are becoming more common. Although mifepristone is the preferred drug used to initiate the abortion in Europe, parts of Asia and in the US, it is not available in many parts of the world such as Canada, South America and most of Africa. While methotrexate is an acceptable and more widely available alternative, concerns about the safety of administration have discouraged some providers from using it. The cost of either mifepristone or methotrexate may also be barriers to widespread use. Misoprostol is inexpensive and easily available and is used alone for abortion both by the women themselves and by medical providers. Effective use of a single safe medication will reduce the number of medications women are exposed to.

Reported effectiveness rates for misoprostol alone in terminating pregnancies less than 8 weeks range from 64 to 94%, with varying doses and protocols. Use of misoprostol in early pregnancy is associated with an increased risk of Mobius syndrome in infants. For this reason, it is important that the most effective regimen is used for abortion to prevent failures.

A summary of the published protocols and results are as follows. A rate of 91.3% was found using 800 mcg vaginally every 24 hours for three doses, with higher effectiveness before 42 days gestation. A dose of 400 mcg sublingual misoprostol repeated every 24 hours for three doses resulted in 86% success. When mifepristone followed by 400 mcg misoprostol orally was compared to 800 mcg misoprostol vaginally, the effectiveness rate of the misoprostol alone was 88% and there were more prostaglandin side effects compared to the combined drug regimen. These side effects were reduced with prophylactic acetominophen and loperamide. Another centre reported a 90.8% effectiveness rate with two doses of 800 mcg misoprostol vaginally. One study assessed women after each dose of 800 mcg vaginal misoprostol and found that only 71.8% aborted after one dose and 92.1% aborted after multiple doses. When 800 mcg vaginally was repeated every 48 hours for three doses, an effectiveness rate of 93.6% was obtained. The same rate was obtained using 1000 mcg. When only 600 mcg vaginally was used, the effectiveness rate was only 64% repeating the dose every 8 hours did not improve the effectiveness. Similar rates were found for adolescents.

One proposed hypothesis for the 64-94% range in effectiveness between these various protocols is that sublingual misoprostol has a higher peak serum concentration than oral or vaginal misoprostol. In other words, the mean time to peak concentration for sublingual misoprostol is similar to oral misoprostol at 26 minutes and the area under the MPA curve is similar to moistened vaginal misoprostol.

The regimen planned for this study is a one-step procedure reported at the International Consortium for Medical Abortion meeting in Johannesburg, October 2004 by Iheoni Obineche. He reported a series of 80 cases in which 79 (98.8%) aborted within 12 hours of receiving 400 mcg vaginal misoprostol after a thorough vaginal cleanse plus 400 mcg sublingual misoprostol administered at the same time. This will be compared to the standard protocol based on the National Abortion Federation and SOGC which is 50mg/m2 of methotrexate injected intramuscularly followed by misoprostol 800mcg per vaginal 4-7 days later.

Rationale:

In countries where abortion is illegal and common such as those in Africa and South America, it is important to find a regimen using misoprostol alone which has a higher completion rate than those regimens usually used.

Trial Objectives:

The primary objective of this study is to determine if misoprostol alone using this regimen is as effective as the investigators' current practice of methotrexate followed by misoprostol for early abortion. The secondary objectives are to compare side effects and to assess acceptability.

Study Design and Duration:

This is a randomized controlled open-label trial. Women requesting medical termination of pregnancy at 7 weeks gestation or less will be recruited.

The study protocol, risks, benefits, visit schedule and consent will be reviewed with each potential subject. The informed consent will include the statement "if the treatment does not work, I have been advised to agree to a surgical abortion". A haemoglobin and Rh factor will be obtained and reviewed. A focussed history and physical examination will be performed. Gestational dating will be done by endovaginal ultrasound using the following criteria: gestational age (days) = mean sac diameter (mm) + 30 or embryonic pole (mm) + 42. Mean sac diameter is used only if there is no embryonic pole. This method has been described by Rossavik and Goldstein.

Randomization will be performed by using a computer generated list of block random numbers and sealed, numbered, opaque envelopes will be prepared by a staff member not involved in the information/consent process.

In both groups, women who are Rh negative will receive 120 :g Rh(D) immune globulin on Day 1. The methotrexate/misoprostol group will be given 50 mg/m2 methotrexate and both written and oral instructions. At least 72 hours after the methotrexate (Day 4-7), they will be asked to moisten four 200 :g tablets of misoprostol with a few drops of water each and insert them into the vagina. On Day 1, the misoprostol-only group will receive 400 :g misoprostol sublingually and the doctor will use a speculum and warm water to cleanse the vagina, moisten 400 :g misoprostol with warm water and place it in the vaginal fornices. All women will also be given six tablets of acetaminophen with codeine, two tablets of diphenhydramine, and six tablets of 400 mg ibuprofen to use for side effects.

All subjects will return to the office within 7 days of having the misoprostol and have another vaginal ultrasound. If they have not aborted, they will be offered three options; waiting, using additional doses of misoprostol or surgery. If the abortion is failed as evidenced by embryonic cardiac activity on Day 15, these women will be scheduled for surgical aspiration. At the first follow-up visit, information will be obtained about completion of the abortion, and then about the woman's experience of bleeding, pain and side effects. Pain will be measured by an 11-point numeric pain scale, using the question "On a scale of 0 to 10, where 0 is no pain and 10 is pain as bad as it can be, what was the worst pain like for you?". They will be asked, "If you were in the same situation, would you choose a medical or surgical abortion? If given the choice, would you choose the same medications you received in this study?". These scales and questions have been reported in other studies.

The main outcome measure is effectiveness after the first dose of misoprostol measured by the number of abortions completed at the first follow-up visit. The investigators will also compare the rate of surgery, the time taken to abort (based on history), side effects, pain and satisfaction. Previous studies have had about 86% of women prefer a medical abortion, 39.2% had nausea, 24.8% had vomiting, 25.9% had fever, 27.2% had headache, 41.8% had chills, and 39.8% had fatigue. The investigators do not expect the side effects to be substantially different. Previously the mean pain scores were 6.3 on an 11-point pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Request for elective abortion
* Ability to understand the consent form
* A pregnancy of 7 weeks gestation or less on Day 1
* Documented by endovaginal ultrasound
* Willingness to comply with visit schedules

Exclusion Criteria:

* Haemoglobin less than 90 g/L
* Uncontrolled seizure disorder
* Active liver disease (aspartate aminotransferase >2x normal)
* Renal insufficiency (serum creatinine >120umol/L)
* A history of intolerance to methotrexate or misoprostol

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2005-09 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
completion of abortion by first follow-up visit

SECONDARY OUTCOMES:
surgery rate
side effects
acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Wiebe, MD, Principal Investigator — UBC
Locations (1):
- Wiebe Early Abortion Clinic, Vancouver, British Columbia, Canada